CLINICAL TRIAL: NCT00339066
Title: Treatment Outcomes of Vascular Depression
Brief Title: Effect of Brain Lesion Severity on Treatment Response in Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2524; R01MH062158 (NIH); DATR A4-GPX
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2008-02

CONDITIONS: Depression
Keywords: Late-Life Depression
MeSH Terms: conditions — Depression | interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline

SUMMARY:
This study will determine the relationship between brain lesion severity, treatment response, and frontal lobe brain function in people with late-life depression (LLD).

DETAILED DESCRIPTION:
Depression in older adults is a major public health problem and it often goes underdiagnosed and undertreated. A significant number of people with LLD, especially those with cerebrovascular risk factors, have subcortical grey matter and frontal deep white matter brain lesions. Some studies suggest that these lesions, or hyperintensities, may be associated with poor acute and long-term depression treatment response. Similarly, studies have shown that people with LLD frequently have functional deficits in the frontal lobe portion of their brains. This dysfunction has been shown to be associated with poor acute treatment response with a tricyclic antidepressant drug, as well as with a greater risk for depression relapse. The applicability of these findings to other classes of antidepressant medications, such as selective serotonin reuptake inhibitors (SSRIs), however, remains unknown. Additionally, more information is needed about the interaction between frontal brain lesions and executive function deficits in LLD. This study will determine the relationship between brain lesion severity, treatment response, and frontal lobe function in people with late-life depression who are being treated with the SSRI sertraline.

Participants in this open label study will first undergo neuropsychological testing to determine eligibility. All eligible participants will be treated with sertraline for 12 weeks. Dosages will begin at 25 mg per day, and will be increased to 50 mg per day after 4 days. Any other dosage modifications will depend on the participant's individual response to the medication. All participants will have an MRI scan at some point during the study. Assessments of symptoms and treatment response will occur at the study site biweekly until Week 8, and then again at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV of major depressive disorder (MDD)
* Score of greater than 20 on the MADRS (score of greater than 17 for atypical depression)
* Score of greater than 20 on the Mini Mental State Examination (MMSE)

Exclusion Criteria:

* Any condition that may make having an MRI medically inadvisable
* Any severe or unstable medical conditions
* Any known primary neurological disorders, including history of stroke
* Any other simultaneous Axis I disorder
* History of substance or alcohol abuse disorder within 6 months prior to study entry
* Currently at risk for suicide
* History of failed prior adequate trials of two antidepressants for the current depressive episode
* History of failed prior adequate trial of sertraline
* Current use of any other psychoactive medications (medication washout will be required)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2001-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Measured at Week 12: Montgomery-Asberg Depression Scale (MADRS)

SECONDARY OUTCOMES:
Measured at Week 12: Hamilton Depression Rating Scale (Ham-D)
Clinical Global Impression (CGI)
Quality of Life Assessment
Disability Assessment

CONTACTS AND LOCATIONS:
Overall Officials: P. Murali Doraiswamy, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Taylor WD, Kuchibhatla M, Payne ME, Macfall JR, Sheline YI, Krishnan KR, Doraiswamy PM. Frontal white matter anisotropy and antidepressant remission in late-life depression. PLoS One. 2008 Sep 24;3(9):e3267. doi: 10.1371/journal.pone.0003267. PMID 18813343